CLINICAL TRIAL: NCT05894590
Title: Cohort Survey on Non-Acute Safety in Persons With Underlying Diseases Who Are Considered to Be at High Risk of Severe COVID-19 by Using Vaccination Information
Brief Title: Post-Marketing Non-Acute Safety Study in Japan After Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) mRNA-1273 COVID-19 Vaccine in Persons at High Risk of Severe COVID-19
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P917
Record Dates: First submitted 2023-06-06; First posted 2023-06-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants received 2 doses of mRNA-1273 vaccine approximately 4 weeks apart.

SUMMARY:
The goal of this study is to assess serious adverse events associated with hospitalizations in the non-acute phase after vaccination with the mRNA-1273 vaccine in persons with underlying diseases who are considered to have a high risk of severe exacerbation of COVID-19.

DETAILED DESCRIPTION:
Data collected from the JMDC Claims database from May 2020 to October 2022.

ELIGIBILITY:
Inclusion Criteria:

* Participants registered to receive the mRNA-1273 vaccine in the Pep Up vaccination history Database
* Participants who have a history of vaccination with the mRNA-1273 vaccine in the Pep-Up vaccination history Database and the observation start date is at least 6 months prior to vaccination with the mRNA-1273 vaccine and have underlying diseases.

Exclusion Criteria:

* Underlying diseases that were determined undetectable by the pre-screening of JMDC
* Participants who did not consent to the questionnaire.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was selected from participants who were registered to receive the mRNA-1273 vaccine in the Pep Up vaccination history Database whose start date of observation in the claim database was within 6 months or more before vaccination with mRNA-1273 vaccine, and those who met the definition of underlying disease based on the claim data for 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 13680 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Serious Events Associated With all-Cause Hospitalizations | Up to 1 year post vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- CMIC Co., Ltd, Tokyo, Japan